CLINICAL TRIAL: NCT02901132
Title: Association Between Different Parameters of Nutritional Assessment and Clinical Outcomes in Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, PHD, Federal University of Minas Gerais
Other Study IDs: FUMinas Gerais
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Cancer; Postoperative Complications; Sarcopenia
MeSH Terms: conditions — Neoplasms; Postoperative Complications; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of abdominal rectal muscles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer group 1: Colorectal cancer patients, under 18 years old, no inflammatory disease, weight loss greater 10% habitual body weight, sarcopenic.
- Control group: No cancer patients, under 18 years old, no inflammatory disease, no weight loss, no sarcopenic.

SUMMARY:
Malnutrition in oncologic patients has a negative impact on post- surgical recovery, survival and quality of life. The etiology of malnutrition in cancer patients is multifactorial, therefore, the nutritional assessment should be carried out by different parameters. The objective of this study is to investigate the association and prognostic value of five distinct methods of nutritional assessment (molecular, body composition, functional, anthropometric and subjective) in relation to postoperative complications and short-term survival in patients with cancer. Regarding the molecular parameter, mtor signaling pathwayon will be assessed in rectus muscle samples, harvested in the moment of the operation. Body composition was assessed by computed tomography (CT) and bioelectrical impedance test was conducted to evaluate the phase angle. Handgrip strength was used to determine functionality. The percentage of weight loss in relation to usual weight was the anthropometric parameter used. Subjective Global Assessment (SGA) was used to provide the nutritional diagnosis. Postoperative complications were classified according to the Dindo and Clavien classification. Overall time survival was the period between the first assessment of the patients until death or end of follow-up. Chi-square test, t test, Kaplan-Meier method and the Log Rank test and regression analysis will be used (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic cancer confirmed
* Over 18 years old
* Accepted the terms of survey

Exclusion Criteria:

* Tumor synchronic
* Inflamattory disease
* Under 18 years old
* No accepted the terms of survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients that will be submitted a surgical treatment at University Hospital of University Federal of Minas Gerais.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | August, 2016
  According to the Dindo-Clavien protocol

SECONDARY OUTCOMES:
Survival | July, 2016
  Follow up using medical records and telephone contacts

OTHER OUTCOMES:
mtor signaling pathway | December, 2016
  mTOR Elisa kits

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - UFMG Hospital, Belo Horizonte, Minas Gerais
  - Hospital of Clinics of the University Federal of Minas Gerais, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: Yes
Scientific publications

REFERENCES:
- [Derived] Mauricio SF, Xiao J, Prado CM, Gonzalez MC, Correia MITD. Different nutritional assessment tools as predictors of postoperative complications in patients undergoing colorectal cancer resection. Clin Nutr. 2018 Oct;37(5):1505-1511. doi: 10.1016/j.clnu.2017.08.026. Epub 2017 Sep 4. PMID 28918167